CLINICAL TRIAL: NCT06373211
Title: Early Immunotherapy with Intravenous Immunoglobulin, Cyclophosphamide and Methylprednisolone in Patients with Anti-Hu-associated Paraneoplastic Sensory Neuronopathy
Acronym: NESPA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP230701; 2023-506942-22-01 (Other: CTIS)
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Paraneoplastic Sensory Neuronopathy
Keywords: Sensory neuronopathy; Paraneoplastic syndrome; Early immunotherapy
MeSH Terms: conditions — Paraneoplastic Syndromes | interventions — gamma-Globulins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Early immunotherapy (Experimental): Early immunotherapy with intravenous immunoglobulin, cyclophosphamide and methylprednisolone
  Interventions: Drug: Immunoglobulins IV (CLAYRIG); Drug: Cyclophosphamide IV; Drug: Methylprednisolone IV

INTERVENTIONS:
Drug: Immunoglobulins IV (CLAYRIG) — Patients will be treated with cycles of :
  - Intravenous (IV) immunoglobulins: 2 g/kg per cycle, over 3 to 5 days (D1 to D3 or D5).
  Cycles will be administered every 4 weeks for a total of 3 first cycles
Drug: Cyclophosphamide IV — Patients will be treated with cycles of :
  - Cyclophosphamide IV: 1 g on the first day (D1). Cycles will be administered every 4 weeks for a total of 6 cycles
Drug: Methylprednisolone IV — Patients will be treated with cycles of :
  Methylprednisolone IV: 1 g/day for 3 days (D1 to D3). Cycles will be administered every 4 weeks for a total of 6 cycles

SUMMARY:
Paraneoplastic Neurological Syndromes are rare autoimmune complications linked to the presence of systemic cancer. Despite their autoimmune origin, they have historically shown little response to immunotherapy. The reason for this failure is probably related to too late administration of immunotherapy, at a stage where the inflammation has already disappeared and irreversible neuronal loss has occurred. The protocol focuses on patients with anti-Hu antibody sensory neuronopathy. This single arm trial consists of an early immunotherapy combining Intravenous Immunoglobulin (IVIG) for 3 months, cyclophosphamide and methylprednisolone for 6 months, at the rate of 1 cycle per month. The percentage of patients with clinical improvement will be evaluated (ONLS) at 3 months. The tolerance of the treatment will also be evaluated as well as other functional scales at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* "Possible" sensory neuronopathy according to the criteria of Camdessanché et al. [2] with ONLS score ≥ 1
* Dominant picture of sensory ataxia (damage to the central nervous system and/or the neuromuscular junction is allowed, provided that it has a minor impact on the patient's disability)
* Positive anti-Hu antibodies in blood and/or cerebrospinal fluid
* Outpatient (modified Rankin Score (mRS) 2 or 3)
* Onset of neurological symptoms less than 3 months ago
* Free, informed, written and signed consent
* Affiliation to a social security or beneficiary scheme (except AME)

Exclusion Criteria:

* Known hypersensitivity to one of the treatments under study, to their metabolites, or to one of the excipients
* Absolute contraindications to IVIg: selective IgA deficiency, known thrombophilia, patients suffering from type I or II hyperprolinemia, hypersensitivity to human immunoglobulins
* Absolute contraindications to cyclophosphamide: vaccination against yellow fever in the 3 months preceding inclusion, acute urinary infection, pre-existing hemorrhagic cystitis, urinary tract obstruction, acute bone marrow failure
* Contraindication to methylprednisolone: live vaccines, or live attenuated vaccines within 3 months, infectious state or evolving virus (hepatitis, herpes, chickenpox, shingles)
* More than two courses of IVIg administered within 3 months before recruitment
* Other concomitant immunotherapy
* Other cause of immunosuppression (acquired or congenital)
* Treatment with checkpoint inhibitors in progress or completed less than 3 months previously
* Woman or man without effective contraception
* Pregnant or breastfeeding woman
* History of psychiatric or general illnesses that may contraindicate treatment
* Patients unable to complete the follow-up required by the study
* Patients under guardianship or curatorship
* Patient deprived of liberty by a judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with clinical improvement on the ONLS (Overall Neuropathy Limitations Scale) at 3 months | At 3 months

SECONDARY OUTCOMES:
Percentage of patients with clinical improvement on the ONLS (Overall Neuropathy Limitations Scale) at 3 and 6 months | At 3 months and at 6 months
Percentage of patients with improvement in the ataxic component on the Score of Ataxia scale at 3 and 6 months | At 3 months and at 6 months
Percentage of patients with improvement in neuropathic pain on the Numeric Rating Scale (NRS) at 3 and 6 months | At 3 months and at 6 months
Percentage of patients with functional improvement on the modified Rankin Score (mRS) at 3 and 6 months | At 3 months and at 6 months
Percentage of patients with functional improvement on the Barthel Index (BI) at 3 and 6 months | At 3 months and at 6 months
Percentage of patients alive and without tumor progression at 6 months | At 6 months
Tolerance to treatment | Through study completion, a maximum of 36 months
  Will be assessed by the frequency and severity of expected and unexpected adverse effects recorded during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Psimaras, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.